CLINICAL TRIAL: NCT03616691
Title: A Phase II Single-arm Trial of Atezolizumab Monotherapy and Consequent Therapy With Atezolizumab Plus Bevacizumab in Patients With Non-Small Cell Lung Cancer After Failure With Platinum-Containing Chemotherapy
Brief Title: Atezolizumab Monotherapy and Consequent Therapy With Atezolizumab Plus Bevacizumab for NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-05-170
Record Dates: First submitted 2018-07-18; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atezolizumab (Experimental): The dose level of atezolizumab proposed to be tested in this study is 1200 mg administered by IV infusion every 3 weeks (q3w)
  Interventions: Drug: Atezolizumab
- Atezolimab+Bevacizumab (Experimental): Once radiologic progression confirmed from atezolizumab monotherapy (stage 1), 1200mg of atezolizumab would be administered with 15mg/kg of bevacizumab as combination therapy (stage 2). Both of drugs are administered via intravenous infusion every 3 weeks.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Stage I: The dose level of atezolizumab proposed to be tested in this study is 1200 mg administered by IV infusion every 3 weeks (q3w)
Drug: Bevacizumab — Stage II: Once radiologic progression confirmed from atezolizumab monotherapy (stage 1), 1200mg of atezolizumab would be administered with 15mg/kg of bevacizumab as combination therapy every 3 weeks.
  Other Names: Atezolizumab
  Arms: Atezolimab+Bevacizumab

SUMMARY:
This is a single-arm phase II trial to evaluate the efficacy and safety of atezolizumab and bevacizumab combination therapy (stage 2) after radiologic progression of atezolizumab monotherapy (stage 1) in Korean patients with locally advanced or metastatic NSCLC who have progressed during or following a platinum-containing regimen. Initially, patients will be treated with Atezolizumab 1200mg every 3 weeks as a single agent (stage 1). After radiologic progression from atezolizumab monotherapy, patients will be consequently treated with atezolizumab (1200mg every 3 weeks) and combination with bevacizumab (15mg/kg every 3 weeks). Exploratory biomarkers will be observed in order to identify predictive biomarkers correlated to response and to evaluate the changes of local and systemic immune profile between baseline and at the time of progression.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for study entry:

1. Signed Informed Consent Form
2. Ability to comply with protocol
3. 20 years old or older
4. Histologically confirmed stage IIIb, IV or recurrent non-squamous cell NSCLC
5. Baseline and repeat biopsy at the time of progression is mandatory. Repeat biopsy at progression to atezolizumab with bevacizumab is optional.
6. Disease progression during or following treatment with a prior platinum-containing regimen for locally advanced, unresectable/inoperable or metastatic NSCLC or disease recurrence within 6 months of treatment with a platinum-based adjuvant/neoadjuvant regimen or combined modality (e.g.,chemoradiation) regimen with curative intent.
7. ECOG performance status of 0 to 1
8. At least one measurable lesion by RECIST v1.1
9. Patients with brain metastasis may be enrolled provided they are asymptomatic requiring no treatment, or are asymptomatic following therapy such as surgery, WBRT or SRT.
10. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment:

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry.

1. Prior treatment with anti-PD1 or anti-PDL1 inhibitors
2. Patients with a known hypersensitivity to atezolizumab and/or bevacizumab or any of the excipients.
3. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
4. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells.
5. Patients with a sensitizing EGFR mutation
6. Patients with a previously detected ALK fusion oncogene
7. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
8. Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease
9. Evidence of interstitial lung disease or active, non-infectious pneumonitis
10. Has received a live vaccine within 30 days prior to the first dose of trial treatment
11. Has a known history of Human Immunodeficieny Virus (HIV)
12. Has known active Hepatitis B (e.g. HBsAg reactive) or Hepatitis C (e.g. HCV RNA is detected)
13. Surgery undertaken less than 4 weeks before the study
14. Localized radiotherapy unless completed more than 2 weeks before the study
15. Uncontrolled systemic illness such as DM, CHF, unstable angina, hypertension or arrhythmia
16. Pregnant or breastfeeding or lactating female patients
17. Female participants of childbearing potential will not agree to use to highly effective form(s) of contraception (i.e., one that results in a low failure rate [<1% per year] when used consistently and correctly) during the treatment period and to continue its use for 5 months after the last dose of Atezolizumab
18. Uncontrolled symptomatic brain metastasis
19. Prior history of malignancy within 5 years from study entry except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer, well-treated thyroid cancer
20. Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg) Anti-hypertensive therapy to achieve these parameters is allowable.
21. Prior history of hypertensive crisis or hypertensive encephalopathy
22. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to randomization
23. History of hemoptysis (>,=one-half teaspoon of bright red blood per episode) within 1 month prior to randomization
24. Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
25. Current or recent (within 10 days of Atezolizumab administration use of aspirin (>325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol
26. Current use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes that has not been stable for >2 weeks prior to randomization
27. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to the first dose of bevacizumab
28. History of abdominal or tracheosphageal fistula or gastrointestinal perforation within 6 months prior to randomization
29. Clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
30. Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
31. Serious, non-healing wound, active ulcer, or untreated bone fracture
32. Proteinuria, as demonstrated by urine dipstick or >1.0 g of protein in a 24-hour urine collection All patients with >, =2+ protein on dipstick urinalysis at baseline must undergo a 24 hour urine collection and must demonstrate > 1 g of protein in 24 hours.
33. Clear tumor infiltration into the thoracic great vessels is seen on imaging
34. Clear cavitation of pulmonary lesions is seen on imaging

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary objective for this study is to evaluate efficacy of atezolizumab with bevacizumab after radiologically progress of atezolizumab monotherapy | about 36 months
  measured by disease control rate (DCR) per investigator using RECIST v1.1

SECONDARY OUTCOMES:
Best overall response rate | about 36 months
  Best overall response rate
Progression-free survival | about 36 months
  PFS, defined as the time from the first administration of atezolizumab and bevacizumab to the first occurrence of disease progression as determined by investigator using RECIST v1.1 or death from any cause, whichever comes first
Duration of response | about 36 months
  DOR, defined as the time from first occurrence of a documented objective response to the time of disease progression as determined by the investigator using RECIST v1.1 or death from any cause, whichever comes first
Overall survival | about 36 months
  OS, defined as the time from the first administration of atezolizumab and bevacizumab to death from any cause
Adverse events (AEs) | about 36 months
  Adverse events will be measured by the CTCAE scale, version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, PhD, Principal Investigator — Samsung Medical Center

IPD SHARING:
Plan to Share IPD: No